CLINICAL TRIAL: NCT06840262
Title: Targeted Muscle Reinnervation (TMR) Versus Regenerative Peripheral Nerve Interfaces (RPNI) Versus the Combined Technique of TMR-RPNI to Reduce Chronic and Phantom Limb Pain in Oncologic Amputees: A Randomized Control Pilot Study
Brief Title: Target Muscle Re-innervation and Regenerative Peripheral Nerve Interfaces Alone and in Combination for the Treatment of Residual and Phantom Limb Pain in Cancer Patients Who Have Received an Amputation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0971; NCI-2021-08488 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (targeted muscle reinnervation) (Active Comparator): Patients undergo TMR procedure.
  Interventions: Other: Questionnaire Administration; Procedure: Targeted Muscle Reinnervation
- Arm 2 (regenerative peripheral nerve interface) (Active Comparator): Patients undergo RPNI procedure.
  Interventions: Other: Questionnaire Administration; Procedure: Regenerative Peripheral Nerve Interface Surgery
- Arm 3 (TMI + RPNI) (Experimental): Patients undergo TMR in combination with RPNI.
  Interventions: Other: Questionnaire Administration; Procedure: Regenerative Peripheral Nerve Interface Surgery; Procedure: Targeted Muscle Reinnervation

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Procedure: Regenerative Peripheral Nerve Interface Surgery — Undergo regenerative peripheral nerve interface surgery
  Other Names: Regenerative Peripheral Nerve Interface; RPNI
  Arms: Arm 2 (regenerative peripheral nerve interface); Arm 3 (TMI + RPNI)
Procedure: Targeted Muscle Reinnervation — Undergo targeted muscle reinnervation
  Other Names: TMR
  Arms: Arm 1 (targeted muscle reinnervation); Arm 3 (TMI + RPNI)

SUMMARY:
This clinical trial evaluates two surgical techniques (targeted muscle re-innervation [TMR] and regenerative peripheral nerve interfaces [RPNI]) alone and in combination for the alleviation of chronic residual limb and phantom limb pain in cancer patients who have had an amputation. Chronic residual limb pain and phantom limb pain are debilitating outcomes of traumatic and oncologic amputation. Emerging microsurgical treatments for post-amputation pain are very promising. TMR and RPNI are both approved surgical techniques that involve connecting cut nerves to parts of the muscle as a way to heal and protect the nerves. This trial evaluates these techniques alone and in combination for the treatment of residual and phantom limb pain in cancer patients who have received an amputation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

Determine the relative effectiveness of three surgical techniques, TMR, RPNI, and TMR with RPNI, on chronic and phantom limb pain in the oncologic amputee using the validated Numerical Rating Scale (NRS) and Patient-Reported Outcomes Measurement Information System (PROMIS) Behavior, Intensity, Interference, and Global Health Forms.

SECONDARY OBJECTIVES:

I. To estimate the rate and total quantity of any pain medication use among oncology amputees who received one of the three surgical techniques.

II. To estimate the rate of prosthetic use among oncologic amputees. III. To compare NRS and PROMIS among three surgical techniques to calculate the effect size and project the sample size which will be used to plan a multi-institutional study.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM 1: Patients undergo TMR procedure.

ARM 2: Patients undergo RPNI procedure.

ARM 3: Patients undergo TMR in combination with RPNI.

After completion of study procedure, patients are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 18 years of age who are receiving an amputation for oncologic reasons
* Patients with available mixed major nerves and donor motor nerves in the amputation stump or reconstructive tissue
* Patients able to complete informed consent

Exclusion Criteria:

* Patients under 18 years of age
* Patients unable to give consent
* Patients receiving an amputation for non-oncologic purposes
* Patients with amputations performed for immediate palliation (life expectancy less than 3 months), as this technique takes a minimum of 3-6 months for effect
* Patients with multiple limb amputations
* Patients receiving nerve management in a delayed fashion (patients who have previously received an amputation and present with neuroma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Margaret S Roubaud, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org